CLINICAL TRIAL: NCT07383987
Title: Investigation of Genital Hygiene, Toilet Behaviors, Body Awareness, and Lower Urinary Tract Symptoms in Normal Weight and Overweight/Obese Women
Brief Title: Genital Hygiene, Toilet Behaviors, and LUTS in Normal Weight and Obese Women
Acronym: GH-TB-BA-LUTS
Status: Recruiting | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Özge Çoban, Assistant Professor, Gulhane School of Medicine
Other Study IDs: 2025-035
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Lower Urinary Tract Symptoms (LUTS); Genital Hygiene; Obesity; Toilet Training; Body Awareness; Overweight
Keywords: obesity; lower urinary tract symptoms; toileting behaviour; genital hygiene behaviours; body awareness
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Weight Group: Normal Weight Group: This group consists of female participants aged 18-45 years with a Body Mass Index (BMI) ranging from 18.5 to 24.9 kg/m². These individuals serve as the control group to evaluate baseline genital hygiene habits, toilet behaviors, body awareness, and lower urinary tract symptoms.
- Overweight Group: Overweight Group: This group consists of female participants aged 18-45 years with a Body Mass Index (BMI) ranging from 25.0 to 29.9 kg/m². This group is evaluated to determine the specific impact of being overweight on urogenital health and behavioral factors compared to normal-weight and obese individuals.
- Obese Group: Obese Group: This group consists of female participants aged 18-45 years with a Body Mass Index (BMI) of 30.0 kg/m² or higher. This group is evaluated to investigate how obesity correlates with the severity of lower urinary tract symptoms, genital hygiene practices, and body awareness levels.

SUMMARY:
The aim of this study is to evaluate and compare genital hygiene habits, toilet behaviors, body awareness levels, and lower urinary tract symptoms (LUTS) in women aged 18-45 years, categorized by Body Mass Index (BMI) as normal weight (BMI = 18.5-24.9 kg/m²) and overweight/obese (BMI ≥ 25 kg/m²). The study seeks to improve social participation and quality of life by increasing awareness regarding obesity, genital hygiene, and urogenital health.

H1: There is a significant difference in lower urinary tract symptoms between BMI groups.

H2: There is a significant difference in genital hygiene behaviors between BMI groups.

H3: There is a significant difference in toilet behaviors between BMI groups. H4: There is a significant difference in body awareness levels between BMI groups.

H5: There is a significant relationship between lower urinary tract symptoms and genital hygiene behavior.

H6: There is a significant relationship between lower urinary tract symptoms and toilet behavior.

H7: There is a significant relationship between lower urinary tract symptoms and body awareness.

H8: There is a significant relationship between genital hygiene behavior and body awareness.

H9: There is a significant relationship between toilet behavior and body awareness.

DETAILED DESCRIPTION:
While existing literature often focuses on single variables, this research adopts a holistic approach. The findings will help clarify the behavioral and awareness-related factors underlying the increased risk of LUTS and infections in overweight/obese women. Ultimately, this study aims to contribute to the development of weight-specific preventive strategies to protect women's urogenital health.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Between the ages of 18 and 45
* Body mass index (BMI) between 18.5-24.9 kg/m² for the normal weight group
* Body mass index (BMI) ≥ 25 kg/m² for the overweight/obese group
* Sufficient cognitive function to answer the questionnaires
* Not having entered menopause

Exclusion Criteria:

* Being pregnant or breastfeeding
* History of bariatric surgery
* History of gynecological or urological surgery/operation
* Diagnosis of lower urinary tract infection or presence of active infection -symptoms
* Presence of any neurological disease
* Presence of any psychiatric disease
* Presence of any oncological disease
* Presence of a communication disorder that would interfere with the questionnaire application

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is limited to female participants because the research focuses on urogenital health parameters specific to female anatomy, including genital hygiene practices, toilet behaviors, and the prevalence of lower urinary tract symptoms (LUTS). The validated scales used in this study, such as the Genital Hygiene Inventory, are specifically designed to evaluate habits and symptoms within the female population. Additionally, the study aims to investigate the impact of Body Mass Index (BMI) on pelvic health and behavioral factors that are physiologically and anatomically distinct in women.
Study Population: The study will be conducted on women of normal weight, overweight, and obese women. Snowball sampling will be used to collect data from women of normal weight and overweight women. Data on obese women will be collected from women who apply to the Ankara Etlik City Hospital General Hospital Obesity Center and are selected based on our criteria.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Bristol Female Lower Urinary Tract Symptoms Questionnaire | Baseline (Single assessment at study enrollment)
  The Bristol Female Lower Urinary Tract Symptoms Questionnaire to assess incontinence and other LUTS, sexual health, and quality of life, has a Cronbach's alpha coefficient of 0.78. In the Turkish version's validity and reliability study conducted by Gökkaya et al., the Cronbach's alpha coefficient was found to be 0.931. The Bristol Female Lower Urinary Tract Symptoms questionnaire consists of 19 questions in 5 subscales: storage (questions 1-4), voiding (questions 5-7), incontinence (questions 8-12), sexual life (questions 13-14), and quality of life (questions 15-19). Questions) and has a Likert-type scoring system ranging from 0 to 3 points for questions 4, 13, 14, 17, and 19, and from 0 to 4 points for the others. A high score indicates increased LUTS severity and a negative impact on quality of life and sexual life.
Genital Hygiene Behaviour Scale | Baseline (Single assessment at study enrollment)
  The Genital Hygiene Practices Scale is a five-point Likert-type scale completed by women themselves, consisting of a total of 23 items and 3 subscales. The subscales of the scale are: 'General Hygiene Habits (first 12 items)', 'Menstrual Hygiene (items 13-20)', and 'Awareness of Abnormal Findings (items 21-23). Scale items are scored numerically from 5 to 1, ranging from 'strongly agree' to 'strongly disagree'. The scale ranges from a minimum score of 23 to a maximum score of 115, with items 7, 14, 19, 20, and 23 being reverse-scored. Higher scores on the scale indicate positive genital hygiene behavior.
Toilet Behaviors - Women's Elimination Behaviors Scale | Baseline (Single assessment at study enrollment)
  The Toilet Behavior-Female Voiding Behavior Scale consists of 18 questions. The Turkish version of the scale consists of 15 questions. The Urination Behavior Scale for Women consists of subgroups such as preferred location for urination (2 items), early urination (4 items), delaying urination (3 items), difficulty urinating (4 items), preferred position for urination (2 items), and each item is scored as 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The internal consistency and reliability of the five subgroups range from 0.70 to 0.88, and the Cronbach's alpha coefficient is 0.81.
Body Awareness Questionnare | Baseline (Single assessment at study enrollment)
  The Body Awareness Questionnaire is an 18-item measure that assesses an individual's reported sensitivity to bodily processes and their ability to predict bodily responses. The Body Awareness Questionnaire has four subscales: 'prediction of bodily responses', 'sleep-wake cycle', 'prediction at the onset of illness', and 'attention to changes and responses in bodily processes', and a 7-point Likert scale is used for evaluation. In this scale, responses are rated from 1 (does not describe me at all) to 7 (describes me completely), and the total score is obtained by adding up the scores for each item. The higher the total score, the higher the body awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Özge ÖZKUTLU, Principal Investigator — Assistant Professor, Department of Physiotherapy and Rehabilitation, Faculty of Physiotherapy and Rehabilitation, University of Health Sciences
Locations (1):
- Etlik City Hospital, Ankara, KEÇİÖREN, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Newman, D.K., et al., Toileting Behaviors and Lower Urinary Tract Symptoms: A Cross-sectional Study of Diverse Women in the United States. Int J Nurs Stud Adv, 2021. 3.
- [Background] Amous, Y., et al., Lower urinary tract symptoms among normal-weight, overweight, and obese palestinians: a study of prevalence and impact on the quality of life. BMC Urol, 2024. 24(1): p. 199.
- [Background] Shang, X., et al., Association of overweight, obesity and risk of urinary incontinence in middle-aged and older women: a meta epidemiology study. 2023. Volume 14 - 2023.
- [Background] Karaca, S. and B. Bayar, TURKISH VERSION OF BODY AWARENESS QUESTIONNAIRE: VALIDITY AND RELIABILITY STUDY. Türk Fizyoterapi ve Rehabilitasyon Dergisi, 2021. 32(1): p. 44-50.
- [Background] Shields, S., M. Mallory, and A. Simon, The Body Awareness Questionnaire: Reliability and Validity. Journal of Personality Assessment - J PERSONAL ASSESS, 1989. 53: p. 802-815.
- [Background] seyhan ak, E., et al., Tuvalet Davranışı-Kadınların Boşaltım Davranışları Ölçeğinin Türkçe'ye Uyarlanması: Geçerlik ve Güvenirlik Çalışması. Turkiye Klinikleri Journal of Nursing Sciences, 2019. 11.
- [Background] Wang, K. and M.H. Palmer, Development and validation of an instrument to assess women's toileting behavior related to urinary elimination: preliminary results. Nurs Res, 2011. 60(3): p. 158-64.
- [Background] Karahan, N., Development of "Genital Hygiene Behaviours Scale": Study of Validity and Reliability. 2017. 18(3): p. 0-0.
- [Background] Khalaf, K.M., et al., Lower urinary tract symptom prevalence and management among patients with multiple sclerosis. Int J MS Care, 2015. 17(1): p. 14-25.
- [Background] Gökkaya, C., et al., Validation of Turkish Version of Bristol Female Lower Urinary Tract Symptom Index. Journal of Clinical and Analytical Medicine, 2012. 3: p. 415-418.
- [Background] Jackson, S., et al., The Bristol Female Lower Urinary Tract Symptoms questionnaire: development and psychometric testing. Br J Urol, 1996. 77(6): p. 805-12.
- See also: Lower urinary tract symptoms among normal-weight, overweight, and obese palestinians: a study of prevalence and impact on the quality of life. — https://doi.org/10.1186/s12894-024-01587-5
- See also: Toileting Behaviors and Lower Urinary Tract Symptoms: A Cross-sectional Study of Diverse Women in the United States — https://doi.org/10.1016/j.ijnsa.2021.100052
- See also: Association of overweight, obesity and risk of urinary incontinence in middle-aged and older women: a meta epidemiology study. 2023. — https://doi.org/10.3389/fendo.2023.1220551